CLINICAL TRIAL: NCT01346293
Title: Safety and Immunogenicity of DTap-IPV (Diphtheria and Tetanus Toxoids and Acellular Pertussis Vaccine Adsorbed Combined With Inactivated Poliovirus Vaccine) Compared to DAPTACEL® (Diphtheria and Tetanus Toxoids and Acellular Pertussis Vaccine Adsorbed) + IPOL® (Poliovirus Vaccine Inactivated) as the 5th Dose in Children 4 to 6 Years of Age
Brief Title: Study of DTap-IPV Compared to DAPTACEL® and IPOL® as the 5th Dose in Children 4 to 6 Years of Age
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: M5I02; U1111-1116-4842 (Other: WHO)
Record Dates: First submitted 2011-04-29; First posted 2011-05-02 (Estimated); Results first posted 2015-05-29 (Estimated); Last update posted 2015-06-03 (Estimated); Status verified 2015-05

CONDITIONS: Tetanus; Diphtheria; Pertussis; Measles; Polio
Keywords: Tetanus; Diphtheria; Pertussis; DTap-IPV; DAPTACEL®; VARIVAX®
MeSH Terms: conditions — Tetanus; Diphtheria; Whooping Cough; Measles; Poliomyelitis | interventions — Tetanus Toxoid; Chickenpox Vaccine; Diphtheria-Tetanus-acellular Pertussis Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Study Group 1 (Experimental): Participants will receive concomitantly a dose of DTap-IPV, a dose of M-M-R®II, and a dose of VARIVAX® vaccine on Day 0
  Interventions: Biological: Diphtheria and Tetanus Toxoids and Acellular Pertussis + Measles, Mumps, Rubella + Varicella Virus
- Study Group 2 (Experimental): Participants will receive concomitantly a dose of DAPTACEL®, a dose of IPOL®, a dose of M-M-R®II, and a dose of VARIVAX® vaccines on Day 0
  Interventions: Biological: Diphtheria and Tetanus Toxoids and Acellular Pertussis + Poliovirus + MMR + Varicella Virus
- Study Group 3 (Experimental): Participants will receive concomitantly a dose of DTap-IPV with or without a dose of M-M-R®II and a dose of VARIVAX® on Day 0
  Interventions: Biological: Diphtheria and Tetanus Toxoids and Acellular Pertussis + Measles, Mumps, Rubella + Varicella Virus
- Study Group 4 (Experimental): Participants will receive concomitantly a dose of DAPTACEL® vaccine, a dose of IPOL® vaccine with or without a dose of M-M-R®II and a dose of VARIVAX® vaccines on Day 0
  Interventions: Biological: Diphtheria and Tetanus Toxoids and Acellular Pertussis + Poliovirus + MMR + Varicella Virus

INTERVENTIONS:
Biological: Diphtheria and Tetanus Toxoids and Acellular Pertussis + Measles, Mumps, Rubella + Varicella Virus — 0.5 mL, Intramuscular (DTap-IPV); Subcutaneous (M-M-R®II and VARIVAX®)
  Other Names: DTap-IPV; M-M-R®II; VARIVAX®
  Arms: Study Group 1
Biological: Diphtheria and Tetanus Toxoids and Acellular Pertussis + Poliovirus + MMR + Varicella Virus — 0.5 mL, Intramuscular (IM) DAPTACEL®; Subcutaneous (SC) MMR®II and VARIVAX®; IM or SC IPOL®
  Other Names: DAPTACEL®; IPOL®; M-M-M R®II; VARIVAX®
  Arms: Study Group 2
Biological: Diphtheria and Tetanus Toxoids and Acellular Pertussis + Measles, Mumps, Rubella + Varicella Virus — 0.5 mL, Intramuscular (DTap-IPV); Subcutaneous (M-M-R®II and VARIVAX®)
  Other Names: DTap-IPV; M-M-R®II; VARIVAX®
  Arms: Study Group 3
Biological: Diphtheria and Tetanus Toxoids and Acellular Pertussis + Poliovirus + MMR + Varicella Virus — 0.5 mL, Intramuscular (IM) DAPTACEL®; Subcutaneous (SC) MMR®II and VARIVAX®; IM or SC IPOL®
  Other Names: DAPTACEL®; IPOL®; M-M-R®II; VARIVAX®
  Arms: Study Group 4

SUMMARY:
The study was designed to compare the safety and immunogenicity of DTap-IPV with DAPTACEL® + IPOL® as the 5th dose booster in children ≥ 4 to < 7 years of age in the US and Puerto Rico who were previously vaccinated with DAPTACEL® and/or Pentacel® vaccines only.

Primary Objectives:

* To compare the pertussis [Pertussis Toxoid (PT), Filamentous Haemagglutinin (FHA), Pertactin (PRN), and Fimbriae Types 2 and 3 (FIM)] booster responses and geometric mean concentrations (GMCs) (as measured by enzyme-linked immunosorbent assay [ELISA]) following DTap-IPV vaccination to those elicited following DAPTACEL® + IPOL® vaccination when administered as a 5th dose.
* To compare the diphtheria and tetanus booster responses and GMCs (as measured by ELISA) following DTap-IPV vaccination with those elicited following DAPTACEL® + IPOL® vaccinations when administered as a 5th dose .
* To compare the Inactivated Poliovirus Vaccine booster responses (as measured by neutralizing assay) following DTap-IPV vaccination with those elicited following DAPTACEL® + IPOL® vaccinations.

Observational Objectives:

* To compare the polio (types 1, 2, and 3) geometric mean titers (GMTs) following DTap-IPV vaccination with those elicited following DAPTACEL® + IPOL® vaccinations.
* To assess the safety of DTap-IPV vaccine or DAPTACEL® + IPOL® vaccine when administered as the fifth dose booster vaccine in participants previously vaccinated with DAPTACEL and/or Pentacel vaccines.

DETAILED DESCRIPTION:
All participants will be randomized to receive either one dose each of DTap-IPV + Measles, Mumps, and Rubella Virus Vaccine Live (M-M-R®II) + VARIVAX® or one dose each of DAPTACEL® + IPOL® + M-M-R®II + VARIVAX® on Day 0.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥ 4 to < 7 years on the day of inclusion
* Informed consent form has been signed and dated by the parent/guardian before the first study-related procedure
* Subject and parent/guardian are able to attend all scheduled visits and to comply with all trial procedures
* Subject has documented completion of primary infant series and booster with DAPTACEL® and/or Pentacel® vaccine(s) only.

Exclusion Criteria:

* Participation in another clinical trial investigating a vaccine, drug, medical device, or medical procedure in the 4 weeks preceding the trial vaccination
* Planned participation in another clinical trial during the present trial period
* Receipt of any vaccine in the 4 weeks preceding the trial vaccination, except for any influenza vaccine, which may be received at least 2 weeks before study vaccines
* Planned receipt of any vaccine in the 4 weeks following the trial vaccination except for any influenza vaccine, which may be received at least 2 weeks after study vaccines
* Receipt of blood or blood-derived products in the past 3 months
* Known or suspected congenital or acquired immunodeficiency; or receipt of immunosuppressive therapy such as anti-cancer chemotherapy or radiation therapy within the preceding 6 months; or long-term systemic corticosteroid therapy (prednisone or equivalent for more than 2 consecutive weeks within the past 3 months)
* History of human immunodeficiency virus (HIV), hepatitis B, or hepatitis C
* History of diphtheria, tetanus, or pertussis infection, confirmed either clinically, serologically, or microbiologically
* Known systemic hypersensitivity to any of the vaccines' components, or history of a life-threatening reaction to the vaccines used in the trial or to a vaccine containing any of the same substances
* Laboratory-confirmed thrombocytopenia, contraindicating intramuscular vaccination
* Bleeding disorder, or receipt of anticoagulants in the 3 weeks preceding inclusion, contraindicating intramuscular vaccination
* Chronic illness that, in the opinion of the Investigator, is at a stage where it might interfere with trial conduct or completion
* Identified as employees of the Investigator or study center, with direct involvement in the proposed study or other studies under the direction of that Investigator or study center, as well as family members (i.e., immediate, husband, wife and their children, adopted or natural) of the employees or the investigator.

Ages: 4 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 3372 (Actual)
Dates: Start 2011-04; Primary Completion 2013-05 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sanofi Pasteur Inc.
Locations (64):
- United States (63):
  - Birmingham, Alabama
  - Pinson, Alabama
  - Trussville, Alabama
  - Chandler, Arizona
  - Scottsdale, Arizona
  - Jonesboro, Arkansas
  - Little Rock, Arkansas
  - La Puente, California
  - Paramount, California
  - Roseville, California
  - Santa Clara, California
  - West Covina, California
  - Longmont, Colorado
  - Thornton, Colorado
  - St. Petersburg, Florida
  - Marietta, Georgia
  - Woodstock, Georgia
  - Indianapolis, Indiana
  - New Albany, Indiana
  - Overland Park, Kansas
  - Topeka, Kansas
  - Crestview Hills, Kentucky
  - Louisville, Kentucky
  - Nicholasville, Kentucky
  - Owensboro, Kentucky
  - Bossier City, Louisiana
  - Haughton, Louisiana
  - Annapolis, Maryland
  - Frederick, Massachusetts
  - Woburn, Massachusetts
  - Bridgeton, Missouri
  - Bellevue, Nebraska
  - Boys Town, Nebraska
  - Lincoln, Nebraska
  - Omaha, Nebraska
  - Brooklyn, New York
  - Fargo, North Dakota
  - Cincinnati, Ohio
  - Fairfield, Ohio
  - Youngstown, Ohio
  - Midwest City, Oklahoma
  - Gresham, Oregon
  - Collegeville, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Scranton, Pennsylvania
  - Bristol, Tennessee
  - Austin, Texas
  - Dallas, Texas
  - Houston, Texas
  - San Antonio, Texas
  - Clinton, Utah
  - Layton, Utah
  - Murray, Utah
  - Orem, Utah
  - Roy, Utah
  - Springville, Utah
  - Syracuse, Utah
  - Burke, Virginia
  - Charlottesville, Virginia
  - Midlothian, Virginia
  - Vienna, Virginia
  - Spokane, Washington
  - Huntington, West Virginia
- San Juan, PR, Puerto Rico

REFERENCES:
- [Derived] Smith MJ, Jordanov E, Sheng X, Tsang PH. Safety and Immunogenicity of DTaP5-IPV Compared With DTaP5 Plus IPV as the Fifth Dose in Children 4-6 Years of Age. Pediatr Infect Dis J. 2017 Mar;36(3):319-325. doi: 10.1097/INF.0000000000001427. PMID 27879555
- See also: Related Info — http://www.sanofipasteur.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study participants were enrolled from 28 April to 16 November 2012 at 70 clinic sites in the United States and Puerto Rico.
Pre-assignment Details: A total of 3372 participants who met all of the inclusion and none of the exclusion criteria were randomized and vaccinated in this study.
Groups:
- DTaP-IPV: Children ≥4 to <7 years of age, who had been previously vaccinated with a 4-dose series of DAPTACEL and/or Pentacel vaccines only, received a single dose of DTaP-IPV intramuscularly
- DAPTACEL®+IPOL®: Children ≥4 to <7 years of age, who had been previously vaccinated with a 4-dose series of DAPTACEL and/or Pentacel vaccines only, received a single dose of DAPTACEL®+IPOL®
Period: Overall Study
Arm/Group | DTaP-IPV | DAPTACEL®+IPOL®
Started | 2743 | 629
Completed | 2676 | 608
Not Completed | 67 | 21
Not completed — Protocol Violation | 30 | 9
Not completed — Lost to Follow-up | 21 | 8
Not completed — Withdrawal by Subject | 15 | 4
Not completed — Other | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | DTaP-IPV | DAPTACEL®+IPOL® | Total
Number analyzed (Participants) | 2743 | 629 | 3372
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 2743 | 629 | 3372
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: Years] | 4.4 (0.5) | 4.4 (0.5) | 4.4 (0.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1330 | 306 | 1636
  Male | 1413 | 323 | 1736
Region of Enrollment [Number; unit: Participants]
  United States | 2743 | 629 | 3372

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Booster Response to the Pertussis Antigens Following Vaccination With Either DTaP-IPV or DAPTACEL® + IPOL® Vaccine
Description: Booster responses to pertussis antigens [pertussis toxoid (PT), filamentous hemagglutinin (FHA), pertactin (PRN), and fimbriae types 2 and 3 (FIM)] were measured by enzyme-linked immunosorbent assay (ELISA). Booster responses were defined as participants with either a pre-vaccination antibody concentration less than lower limit of quantitation (<LLOQ), achieving a post-vaccination level ≥4X LLOQ, or pre-vaccination antibody concentrations ≥LLOQ but <4X LLOQ, achieving a 4-fold rise rate of post-vaccination, or a pre-vaccination antibody concentration ≥4X LLOQ, achieving a 2-fold response.
Time Frame: Day 0 (pre-vaccination) and Day 28 post-vaccination
Population: Anti-pertussis booster responses were assessed in the Per-Protocol Analysis Set.
Measure: Number; unit: Participants
Groups:
- DTaP-IPV: Children ≥4 to <7 years of age, who had been previously vaccinated with a 4 dose series of DAPTACEL and/or Pentacel vaccines only, received a single dose of DTaP-IPV intramuscularly
- DAPTACEL®+IPOL®: Children ≥4 to <7 years of age, who had been previously vaccinated with a 4 dose series of DAPTACEL and/or Pentacel vaccines only, received a single dose of DAPTACEL®+IPOL®
Arm/Group | DTaP-IPV | DAPTACEL®+IPOL®
Number analyzed (Participants) | 263 | 253
Participants
  Anti-Pertussis toxoid (N=252, 247) | 240 | 222
  Anti-Filamentous hemagglutinin (N=255, 248) | 242 | 217
  Anti-Pertactin (N=254, 248) | 246 | 231
  Anti-Fimbriae types 2 and 3 (N=250, 249) | 243 | 230
Statistical Analysis 1: Comparison: DTaP-IPV vs DAPTACEL®+IPOL®; Non-inferiority comparison of post-vaccination anti-pertussis booster response rates in the Per-protocol Analysis Set. The hypothesis was based on testing the difference between 2 proportion parameters; Test type: Non-Inferiority or Equivalence — Non-inferiority of DTaP-IPV was demonstrated if the lower limits of the 2-sided 95% Confidence intervals (CIs) of the difference (DTaP-IPV minus DAPTACEL® + IPOL®) in post-vaccination booster response rates for Anti-Pertussis toxoid antigen between groups were > -10%; Mean Difference (Final Values) = 5.4, 95% CI 2-sided [0.7 to 10.2]
Statistical Analysis 2: Comparison: DTaP-IPV vs DAPTACEL®+IPOL®; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — Non-inferiority of DTaP-IPV was demonstrated if the lower limits of the 2-sided 95% CIs of the difference (DTaP-IPV minus DAPTACEL® + IPOL®) in post-vaccination booster response rates for Anti-Filamentous Haemagglutinin between groups were > -10%; Mean Difference (Final Values) = 7.4, 95% CI 2-sided [2.5 to 21.5]
Statistical Analysis 3: Comparison: DTaP-IPV vs DAPTACEL®+IPOL®; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — Non-inferiority of DTaP-IPV was demonstrated if the lower limits of the 2-sided 95% CIs of the difference (DTaP-IPV minus DAPTACEL® + IPOL®) in post-vaccination booster response rates for the Pertactin antigens between groups were > -10%; Mean Difference (Final Values) = 3.7, 3.7% CI 2-sided [-0.2 to 7.9]
Statistical Analysis 4: Comparison: DTaP-IPV vs DAPTACEL®+IPOL®; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — Non-inferiority of DTaP-IPV was demonstrated if the lower limits of the 2-sided 95% CIs of the difference (DTaP-IPV minus DAPTACEL® + IPOL®) in post-vaccination booster response rates for Fimbriae types 2 and 3 antigens between groups were > -10%; Mean Difference (Final Values) = 4.8, 95% CI 2-sided [0.9 to 9.1]

2. Primary Outcome: Geometric Mean Concentrations of the Pertussis Antibodies Before and Following Vaccination With Either DTaP-IPV or DAPTACEL® + IPOL® Vaccine
Description: Geometric mean concentrations to pertussis antigens (pertussis toxoid [PT], filamentous hemagglutinin [FHA], pertactin [PRN], and fimbriae types 2 and 3 [FIM]) were measured by enzyme-linked immunosorbent assay (ELISA).
Time Frame: Day 0 (pre-vaccination) and Day 28 post-vaccination
Population: Geometric mean concentrations were assessed in the Per-Protocol Analysis Set.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | DTaP-IPV | DAPTACEL®+IPOL®
Number analyzed (Participants) | 263 | 253
Titers
  Anti-PT pre-vaccination (N=254, 248) | 5.16 [4.48 to 5.94] | 4.74 [4.18 to 5.39]
  Anti-PT post-vaccination (N=261, 252) | 121 [108 to 134] | 61.3 [54.5 to 68.9]
  Anti-FHA pre-vaccination (N=255, 248) | 7.93 [6.63 to 9.47] | 9.42 [7.85 to 11.3]
  Anti-FHA post-vaccination (N=263, 253) | 123 [108 to 141] | 79.0 [69.3 to 90.0]
  Anti-PRN pre-vaccination (N=255, 249) | 18.6 [16.2 to 21.3] | 16.7 [14.6 to 19.1]
  Anti-PRN post-vaccination (N=262, 252) | 283 [252 to 317] | 187 [164 to 214]
  Anti-FIM pre-vaccination (N=253, 249) | 31.9 [27.0 to 37.6] | 33.3 [28.3 to 39.2]
  Anti-FIM post-vaccination (N=260, 253) | 506 [448 to 571] | 379 [331 to 433]
Statistical Analysis 1: Comparison: DTaP-IPV vs DAPTACEL®+IPOL®; Hypothesis was based on testing the ratio between the 2 post-vaccination GMCs (GMCQ / GMCD) for each Pertussis antigen and their 2-sided 95% Confidence Intervals; Test type: Non-Inferiority or Equivalence — Non-inferiority of DTaP-IPV was demonstrated if the lower limits of the 2-sided 95% CIs of the ratio (DTaP-IPV / DAPTACEL® + IPOL®) in post-vaccination GMCs for the Pertussis Toxoid antigens between groups were > 2/3; Mean Difference (Final Values) = 1.97, 95% CI 2-sided [1.68 to 2.31]
Statistical Analysis 2: Comparison: DTaP-IPV vs DAPTACEL®+IPOL®; [analysis description as in outcome 2, analysis 1]; Test type: Non-Inferiority or Equivalence — Non-inferiority of DTaP-IPV was demonstrated if the lower limits of the 2-sided 95% CIs of the ratio (DTaP-IPV / DAPTACEL® + IPOL®) in post-vaccination GMCs for the Filamentous Haemagglutinin antigens between groups were > 2/3; Mean Difference (Final Values) = 1.56, 95% CI 2-sided [1.30 to 1.88]
Statistical Analysis 3: Comparison: DTaP-IPV vs DAPTACEL®+IPOL®; [analysis description as in outcome 2, analysis 1]; Test type: Non-Inferiority or Equivalence — Non-inferiority of DTaP-IPV was demonstrated if the lower limits of the 2-sided 95% CIs of the ratio (DTaP-IPV / DAPTACEL® + IPOL®) in post-vaccination GMCs for the Pertactin antigens between groups were > 2/3; Mean Difference (Final Values) = 1.51, 95% CI 2-sided [1.27 to 1.79]
Statistical Analysis 4: Comparison: DTaP-IPV vs DAPTACEL®+IPOL®; [analysis description as in outcome 2, analysis 1]; Test type: Non-Inferiority or Equivalence — Non-inferiority of DTaP-IPV was demonstrated if the lower limits of the 2-sided 95% CIs of the ratio (DTaP-IPV / DAPTACEL® + IPOL® ) in post-vaccination GMCs for the Fimbriae types 2 and 3 antigens between groups were > 2/3; Mean Difference (Final Values) = 1.33, 95% CI 2-sided [1.12 to 1.60]

3. Primary Outcome: Number of Participants With Booster Response to Tetanus and Diphtheria Antigens Following Vaccination With Either DTaP-IPV or DAPTACEL® + IPOL® Vaccine
Description: Anti-Tetanus antibodies were measured by enzyme-linked immunosorbent assay (ELISA). Anti-Diphtheria antibodies were measured by a toxin neutralization test. Booster responses were defined as participants with a pre-vaccination antibody concentration <0.1 IU/ml, achieving a post-vaccination level ≥0.4 IU/ml, or a pre-vaccination antibody concentration ≥0.1 IU/ml but <2.0 IU/ml, achieving a 4-fold rise rate post-vaccination, or a pre-vaccination antibody concentration ≥2.0 IU/ml, achieving a 2-fold response.
Time Frame: Day 0 (pre-vaccination) and Day 28 post-vaccination
Population: Anti-Tetanus and anti-diphtheria booster responses were assessed in the Per-Protocol Analysis Set.
Measure: Number; unit: Participants
Arm/Group | DTaP-IPV | DAPTACEL®+IPOL®
Number analyzed (Participants) | 263 | 253
Participants
  Anti-Tetanus (N=253, 248) | 213 | 209
  Anti-Diphtheria (N=256, 249) | 249 | 247

4. Primary Outcome: Geometric Mean Concentrations of the Tetanus and Diphtheria Antibodies Before and Following Vaccination With Either DTaP-IPV or DAPTACEL® + IPOL® Vaccine
Description: Geometric mean concentrations to anti-tetanus and anti-diphtheria were measured by enzyme-linked immunosorbent assay (ELISA).
Time Frame: Day 0 (pre-vaccination) and Day 28 post-vaccination
Population: Geometric mean concentrations of tetanus and diptheria antibodies were assessed in the Per Protocol Analysis Set.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | DTaP-IPV | DAPTACEL®+IPOL®
Number analyzed (Participants) | 263 | 253
Titers
  Anti-Tetanus pre-vaccination (N=254, 248) | 0.644 [0.548 to 0.758] | 0.608 [0.518 to 0.715]
  Anti-Tetanus post-vaccination (N=262, 253) | 6.42 [5.74 to 7.18] | 5.48 [4.88 to 6.15]
  Anti-Diphtheria pre-vaccination (N=257, 249) | 0.510 [0.437 to 0.596] | 0.426 [0.362 to 0.501]
  Anti-Diphtheria post-vaccination (N=262, 253) | 18.6 [16.6 to 20.8] | 15.5 [13.7 to 17.6]

5. Primary Outcome: Number of Participants With Booster Response to Polio Antigens Following Vaccination With Either DTaP-IPV or DAPTACEL® + IPOL® Vaccine
Description: Anti-poliovirus types 1, 2, and 3 titers were measured by neutralization assay. Booster responses were defined as participants with a pre-vaccination antibody concentration <1:8 dil, achieving a post-vaccination level ≥1:8 dil, or a pre-vaccination antibody concentration ≥1:8 dil, achieving a 4-fold response.
Time Frame: Day 0 (pre-vaccination) and Day 28 post-vaccination
Population: Anti-polio booster responses were assessed in the Per-Protocol Analysis Set.
Measure: Number; unit: Participants
Arm/Group | DTaP-IPV | DAPTACEL®+IPOL®
Number analyzed (Participants) | 263 | 253
Participants
  Anti-Polio 1 (N=249, 248) | 214 | 204
  Anti-Polio 2 (N=249, 248) | 195 | 196
  Anti-Polio 3 (N=247, 248) | 210 | 210

6. Primary Outcome: Geometric Mean Concentrations of Polio Antibodies Before and Following Vaccination With Either DTaP-IPV or DAPTACEL® + IPOL® Vaccine
Description: Geometric mean concentrations to anti-polio were measured by enzyme-linked immunosorbent assay (ELISA).
Time Frame: Day 0 (pre-vaccination) and Day 28 post-vaccination
Population: Geometric mean concentrations of poliovirus antibodies were assessed in the Per-Protocol Analysis Set.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | DTaP-IPV | DAPTACEL®+IPOL®
Number analyzed (Participants) | 263 | 253
Titers
  Anti-Polio 1 pre-vaccination (N=254, 248) | 135 [114 to 160] | 129 [110 to 151]
  Anti-Polio 1 post-vaccination (N=258, 253) | 3477 [3088 to 3915] | 2731 [2384 to 3128]
  Anti-Polio 2 pre-vaccination (N=254, 248) | 214 [183 to 249] | 188 [160 to 221]
  Anti-Polio 2 post-vaccination (N=258, 253) | 3491 [3111 to 3917] | 3894 [3393 to 4468]
  Anti-Polio 3 pre-vaccination (N=252, 248) | 102 [85.1 to 123] | 90.9 [74.5 to 111]
  Anti-Polio 3 post-vaccination (N=258, 252) | 4591 [4011 to 5256] | 3419 [2946 to 3969]

7. Other Pre Specified Outcome: Number of Participants With Seroprotection Against the Tetanus and Diphtheria Antigens Before and Following Vaccination With Either DTaP-IPV or DAPTACEL® + IPOL® Vaccine
Description: Anti-Tetanus antibodies were measured by ELISA. Anti diphtheria antibodies were measured by a toxin neutralization test. Seroprotection for anti-tetanus and anti-diphtheria was defined as antibody concentrations ≥0.1 IU/ml and ≥1.0 IU/ml.
Time Frame: Day 0 (pre-vaccination) and Day 28 post-vaccination
Population: Seroprotection against tetanus and diphtheria antigens was assessed in the Per-Protocol Analysis Set.
Measure: Number; unit: Participants
Arm/Group | DTaP-IPV | DAPTACEL®+IPOL®
Number analyzed (Participants) | 263 | 253
Participants
  Anti-Tetanus pre-vacc. ≥0.1 IU/ml (N=254, 248) | 233 | 221
  Anti-Tetanus pre-vacc. ≥1.0 IU/ml (N=254, 248) | 93 | 89
  Anti-Tetanus post-vacc. ≥0.1 IU/ml (N=262, 253) | 262 | 251
  Anti-Tetanus post-vacc. ≥1.0 IU/ml (N=262, 253) | 259 | 245
  Anti-Diphtheria pre-vacc. ≥0.1 IU/ml (N=257, 249) | 233 | 207
  Anti-Diphtheria pre-vacc. ≥1.0 IU/ml (N=257, 249) | 78 | 72
  Anti-Diphtheria post-vacc. ≥0.1 IU/ml (N=262, 253) | 262 | 252
  Anti-Diphtheria post-vacc. ≥1.0 IU/ml (N=262, 253) | 261 | 252

8. Other Pre Specified Outcome: Number of Participants With Seroprotection Against the Polio Antigens Before and Following Vaccination With Either DTaP-IPV or DAPTACEL® + IPOL® Vaccine
Description: Anti-Poliovirus types 1, 2, and 3 titers were measured by neutralization assay. Seroprotection for anti-polio types was defined as antibody titers ≥1:8 dilution.
Time Frame: Day 0 (pre-vaccination) and Day 28 post-vaccination
Population: Seroprotection (antibody titers ≥1:8 dilution) against polio antigens was assessed in the Per-Protocol Analysis Set.
Measure: Number; unit: Participants
Arm/Group | DTaP-IPV | DAPTACEL®+IPOL®
Number analyzed (Participants) | 263 | 253
Participants
  Anti-Polio 1 pre-vaccination (N=254, 248) | 250 | 245
  Anti-Polio 1 post-vaccinatin (N=258, 253) | 258 | 252
  Anti-Polio 2 pre-vaccination (N=254, 248) | 253 | 247
  Anti-Polio 2 post-vaccination (N=258, 253) | 258 | 253
  Anti-Polio 3 pre-vaccination (N=252, 248) | 244 | 231
  Anti-Polio 3 post-vaccination (N=258, 252) | 258 | 252

9. Other Pre Specified Outcome: Number of Participants With Booster Response to the Polio Antigens Following Vaccination With Inactivated Poliovirus (IPV) Vaccine as a 4th or 5th Dose
Description: Anti-Poliovirus types 1, 2, and 3 titers were measured by neutralization assay. Four-fold rise in booster responses between groups was defined as post/pre-vaccination ≥4.
Time Frame: Day 0 (pre-vaccination) and Day 28 post-vaccination
Population: Booster responses to polio antigens following IPV vaccine as 4th or 5th dose were assessed in the Per-Protocol Analysis Set.
Measure: Number; unit: Participants
Arm/Group | DTaP-IPV | DAPTACEL®+IPOL®
Number analyzed (Participants) | 262 | 252
Participants
  Anti-Polio 1 4th dose (N=238, 235) | 205 | 199
  Anti-Polio 1 5th dose (N=10, 12) | 8 | 4
  Anti-Polio 2 4th dose (N=238, 235) | 188 | 190
  Anti-Polio 2 5th dose (N=10, 12) | 7 | 5
  Anti-Polio 3 4th dose (N=236, 235) | 203 | 202
  Anti-Polio 3 5th dose (N=10, 12) | 6 | 7

10. Other Pre Specified Outcome: Summary of Anti-Polio Geometric Mean Titers in Participants That Received Inactivated Poliovirus (IPV) Vaccine as a 4th and 5th Dose
Description: Anti-Poliovirus types 1, 2, and 3 titers were measured by neutralization assay.
Time Frame: Day 0 (pre-booster vaccination) and Day 28 post-booster vaccination
Population: Anti-Polio geometric mean titers were assessed in the Per-Protocol Analysis Set.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | DTaP-IPV | DAPTACEL®+IPOL®
Number analyzed (Participants) | 263 | 252
Titers
  Anti-Polio 1 pre-4th dose (N=243, 235) | 134 [112 to 159] | 123 [105 to 144]
  Anti-Polio 1 post-4th dose (N=247, 240) | 3471 [3072 to 3921] | 2774 [2420 to 3179]
  Anti-Polio 1 pre-5th dose (N=10, 12) | 194 [70.6 to 533] | 342 [131 to 890]
  Anti-Polio 1 post-5th dose (N=10, 12) | 3327 [1769 to 6256] | 1773 [692 to 4543]
  Anti-Polio 2 pre-4th dose (N=243, 235) | 210 [179 to 246] | 181 [153 to 213]
  Anti-Polio 2 post-4th dose (N=247, 240) | 3495 [3117 to 3920] | 3991 [3470 to 4590]
  Anti-Polio 2 pre-5th dose (N=10, 12) | 274 [135 to 558] | 431 [166 to 1119]
  Anti-Polio 2 post-5th dose (N=10, 12) | 3566 [1205 to 10554] | 2048 [1002 to 4187]
  Anti-Polio 3 pre-4th dose (N=241, 235) | 99.5 [82.1 to 121] | 86.3 [70.6 to 106]
  Anti-Polio 3 post-4th dose (N=247, 239) | 4773 [4168 to 5466] | 3500 [3007 to 4075]
  Anti-Polio 3 pre-5th dose (N=10, 12) | 239 [137 to 417] | 323 [139 to 748]
  Anti-Polio 3 post-5th dose (N=10, 12) | 1663 [687 to 4026] | 2436 [1033 to 5744]

11. Other Pre Specified Outcome: Number of Participants Reporting Solicited Injection-site and Systemic Reactions Following Vaccination With Either DTaP-IPV or DAPTACEL® + IPOL® Vaccine
Description: Solicited injection-site: Pain, Erythema, Swelling, Extensive Swelling of Vaccinated Limb, Change in Limb Circumference. Solicited systemic reactions: Fever (Temperature), Headache, Malaise, and Myalgia. Grade 3 injection-site: Pain, Incapacitating, unable to perform usual activities; Erythema, Swelling, ≥50 mm; Change in limb circumference >50 mm increase over pre-vaccination measurement; Extensive limb swelling (ELS) was considered severe. Grade 3 systemic reactions: Fever ≥39.0˚C; Headache, Malaise, and Myalgia Significant, prevents daily activity.
Time Frame: Day 0 up to Day 28 post-final vaccination
Population: Solicited injection-site and systemic reactions were assessed in the Safety Analysis Set.
Measure: Number; unit: Participants
Arm/Group | DTaP-IPV | DAPTACEL®+IPOL®
Number analyzed (Participants) | 2733 | 621
Participants
  Injection-site Pain (N=2689, 603) | 2081 | 461
  Grade 3 Injection-site Pain (N=2689, 603) | 53 | 18
  Injection-site Erythema (N=2687, 603) | 1587 | 322
  Grade 3 Injection-site Erythema (N=2687, 603) | 484 | 72
  Injection-site Swelling (N=2678, 602) | 1076 | 219
  Grade 3 Injection-site Swelling (N=2678, 602) | 229 | 43
  Extensive limb swelling (N=2666, 598) | 39 | 8
  Grade 3 Extensive limb swelling (N=2666, 598) | 39 | 8
  Change in limb circumference (N=2500, 464) | 1703 | 302
  Grade 3 Change in limb circumference (N=2500, 464) | 4 | 0
  Fever (N=2668, 598) | 161 | 41
  Grade 3 Fever (N=2668, 598) | 35 | 12
  Headache (N=2688, 603) | 419 | 100
  Grade 3 Headache (N=2688, 603) | 15 | 4
  Malaise (N=2687, 603) | 940 | 200
  Grade 3 Malaise (N=2687, 603) | 71 | 20
  Myalgia (N=2688, 603) | 1445 | 317
  Grade 3 Myalgia (N=2688, 603) | 52 | 17

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from Day 0 (post-vaccination) up to Day 28 post-vaccination
Description: The number of participants at risk for each specific solicited injection site and systemic reactions (reported as Other Adverse Events) was based on the number of participants who completed and returned diary cards used for the period.
Arm/Group | DTaP-IPV | DAPTACEL®+IPOL®
Serious Adverse Events (participants affected / at risk) | 21/2733 | 3/621
Other Adverse Events (participants affected / at risk) | 2081/2733 | 461/621
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DTaP-IPV (N=2733) | DAPTACEL®+IPOL® (N=621)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Rectal prolapse (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Immunodeficiency common variable (Immune system disorders) | 1 (1) | 0 (0)
Clostridial infection (Infections and infestations) | 1 (1) | 0 (0)
Croup infectious (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 0 (0)
Lobar pneumonia (Infections and infestations) | 2 (2) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Skull fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Synovitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Autism (Nervous system disorders) | 1 (1) | 0 (0)
Petit mal epilepsy (Nervous system disorders) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 0 (0)
Kawasaki's disease (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5.00% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | DTaP-IPV (N=2733) | DAPTACEL®+IPOL® (N=621)
Injection site induration (General disorders) | 139 (142) | 20 (20)
Cough (Respiratory, thoracic and mediastinal disorders) | 142 (147) | 26 (26)
Injection site Pain (General disorders) | 2081/2689 (2081) | 461/603 (461)
Injection site Erythema (General disorders) | 1587/2687 (1587) | 322/603 (322)
Injection site Swelling (General disorders) | 1076/2678 (1076) | 219/602 (219)
Change in limb circumference (General disorders) | 1703/2500 (1703) | 302/464 (302)
Fever (General disorders) | 161/2668 (161) | 41/598 (41)
Headache (Nervous system disorders) | 419/2688 (419) | 100/603 (100)
Malaise (General disorders) | 940/2687 (940) | 200/603 (200)
Myalgia (Musculoskeletal and connective tissue disorders) | 1445/2688 (1445) | 317 (317)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor must have the opportunity to review at least 60 days prior to submission for publication or presentation. If review indicates that potentially patentable subject matter would be disclosed, publication or public disclosure may be delayed for a maximum of an additional 60 days to allow for filing the necessary patent applications